CLINICAL TRIAL: NCT06289374
Title: The LABS Study: Longitudinal Assessment of Biomarkers After Oesophagogastric Cancer Surgery (BIORESOURCE 2: Longitudinal)
Brief Title: Longitudinal Assessment of Biomarkers After Oesophagogastric Cancer Surgery
Acronym: LABS
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Other Study IDs: 23HH8340
Record Dates: First submitted 2024-02-26; First posted 2024-03-01 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Oesophageal Adenocarcinoma; Gastric Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The LABS study (Bioresource 2: Longitudinal): 200 patients following oesophagogastric cancer resection recruited into BIORESOURCE 1. Following surgery at 3 months, 6 months, 1 year and 2 years: saliva, urine, blood, breath and quality of life questionnaires will be collected.
  Interventions: Other: Biosample collection

INTERVENTIONS:
Other: Biosample collection — Collection of saliva, urine, blood, breath and quality of life questionnaires.

SUMMARY:
Oesophagogastric cancer (cancer of the gullet and stomach) is the fifth most common cancer in England and Wales with 16,000 new cases diagnosed every year. Survival rates are poor with only 15% surviving beyond 5 years. There is also increasing research to understand the cancer biology and factors allowing cancers to progress. It is likely there is a relationship between the cancer-specific microbiome, cells related to inflammation, which promotes cancer progression. The BIORESOURCE 1 study has established a comprehensive resource of matched samples from patients with oesophageal and gastric cancer. This longitudinal study aims to obtain further matched biosamples in the follow-up period after cancer surgery to find biomarkers that may predict treatment response, recurrence and/or long term prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-90 years at the time of initial recruitment
* Gastric/oesophageal adenocarcinoma cohort (biopsy proven adenocarcinoma) recruited into BIORESOURCE 1

Exclusion Criteria:

* Oesophageal squamous cell carcinoma
* Previous oesophageal and gastric resection
* History of another cancer within five years. If a new other cancer type is diagnosed within the sampling time frame, no further samples will be taken.
* Participants with co-morbidities preventing breath collection
* Unable or unwilling to provide informed written consent
* Pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen in a hospital (secondary or tertiary level care) setting
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Salivary microbial biomarkers to predict treatment response and long-term prognosis | 48 months
  Changes in the presence and/or abundance of bacteria over a 2 year period, measured primarily within saliva.

SECONDARY OUTCOMES:
Breath volatile organic compound profile alterations of oesophagogastric cancer pre- and post- treatment | 48 months
  Changes in the VOC profile using gas chromatography mass spectrometry.
Quality of life measure up to 2 years following cancer surgery using validated questionnaires | 48 months
  Assessment in the longitudinal changes of quality of life measures using validated questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No